CLINICAL TRIAL: NCT04397952
Title: Comparison of Two Different Measurement of Endotracheal Tube Cuff Pressure for Ventilatory Associated Pnemonia in Severe Brain Injured Patients
Brief Title: Endotracheal Tube Cuff Pressure Measurement
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017.11.1.02.008.r1.010
Record Dates: First submitted 2020-01-20; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Ventilator Associated Pneumonia; Morality; Trauma, Brain; Endotracheal Aspiration
Keywords: pneumonia, cuff pressure, brain injury
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Brain Injuries, Traumatic; Pneumonia; Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effect of endotracheal cuff pressure measurement technique for preventing ventilatory associated pneumonia.

DETAILED DESCRIPTION:
Aim of this study is to evaluate the effect of endotracheal cuff pressure measurement technique for preventing ventilatory associated pneumonia of severe traumatic brain injured patients in a tertiary level intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

Patients with ASA classification of 1 - 2- 3 patients Patients required mechanical ventilation support for more than 48 hours Patients diagnosed with Traumatic brain injury

Exclusion Criteria:

Official patient relatives who rejected to give informed consent for the study Patients diagnosed with aspiration pneumonia during ICU follow up Patients diagnosed with Acute Respiratory Distress Syndrome Patients diagnosed with cavitary lung lesion Primary lung cancer Metastatic lung cancer Congenitally immune deficiency Leukopenia Neutropenia Tracheostomized patients Post cardiopulmonary arrest patients Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who followed up in a tertiary intensive care unit diagnosed with traumatic brain injury and under mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Duration | 30 days
  Follow up duration in ICU
Ventilation | 30 days
  Mechanically ventilated period
Score | 48.hour - 72.hour - 96.hour
  Clinical Pulmonary Infection Score Change from baseline at 48.hour, 72.hour and 96.hour
CRP | 48.hour - 72.hour - 96.hour
  C Reactive Protein measurement change from Baseline at 48.hour, 72.hour and 96.hour
Oxygenation | 48.hour - 72.hour - 96.hour
  Fractional Inspiratory Oxygen levels change from baseline at 48.hour, 72.hour and 96.hour
PEEP | 48.hour - 72.hour - 96.hour
  Positive End Expiratory Pressure levels change from baseline at 48.hour, 72.hour and 96.hour during ventilatory support

SECONDARY OUTCOMES:
Tracheal aspirate | 0.hour - 48.hour - 72.hour - 96.hour
  Tracheal aspirate sample for culture
Bacterial distribution | 0.hour - 48.hour - 72.hour - 96.hour
  Bacterial distribution of tracheal aspirate culture
Mortality | 30 days
  Total mortality ratio during study period

CONTACTS AND LOCATIONS:
Overall Officials: Salih SS Sevdi, MD, Principal Investigator — Univesity of Health Sciences Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided